CLINICAL TRIAL: NCT03057327
Title: Promoting Early Detection of Melanoma During the Mammography Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Research Professor of Dermatology, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STU00204685
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Melanoma (Skin Cancer)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: sequential single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comparator (Active Comparator): As women exit the changing are they will be asked if they regularly check their skin for concerning moles
  Interventions: Other: Comparator
- Improve awareness of checking moles (Experimental): Posters, brochures, and skin self-examination kits consisting of a ruler, and a lighted magnifying lens will be placed into each of the 8 changing rooms in the mammogram facility.
  Interventions: Behavioral: Improve awareness of checking moles

INTERVENTIONS:
Behavioral: Improve awareness of checking moles — Intervention:
  1. Improve awareness Each of the eight changing rooms will have a large mirror that can be used to see the face and chest. Each room will be equipped with a poster, brochures and the SSE kit consisting of the laminated card with a ruler on one edge and the magnifying lens will be fastened to the wall on a cord.
  2. Provide education The subject may chose to read the poster and a brochure. c) A woman research assistant will perform in-person exit interviews with participants to ascertain if women noticed the poster, and found the information relevant.
  Arms: Improve awareness of checking moles
Other: Comparator — Prior to placing the intervention materials into the changing rooms, 100 eligible subjects will be asked if they regularly check their moles for concerning features. If the response is yes, then they will be asked if they have found concerning moles and what they did next.
  Arms: comparator

SUMMARY:
The proposed study is a pilot and feasibility study designed to develop materials to enhance early detection of melanomas among women at risk to develop melanoma due to indoor tanning, having a family history of melanoma or a personal history of melanoma.

The hypothesis of this study is that women, who are engaged in health promotion by having mammograms, will be able to assess the personal relevance of skin self-examination (SSE), be interested in learning about SSE and able to implement SSE while they are partially disrobed in the privacy of the changing room in the mammogram facility.

DETAILED DESCRIPTION:
After patients complete the mammogram, they return to the changing room and put on their clothing. After exiting the changing room in the Lynn Sage Comprehensive Breast Center of Northwestern Medicine/Prentice Women's Hospital and as they are preparing to leave, a research assistant (RA) will screen potential participants to acquire a randomly selected convenience sample of eligible participants (n=200). The first 100 eligible subjects will be asked if they regularly check their moles for concerning features. If the response is yes, then they will be asked if they have found concerning moles and what they did next. Verbal assent will be obtained.

Then the SSE materials will be placed into the changing rooms and the next 100 eligible subjects will be surveyed. The women, who found the information relevant, will be asked if they chose to check their skin while in the changing room. The skin location checked and use of the SSE kit will be ascertained. Women will be asked if they think they have a concerning mole. If the woman does not find a concerning mole, she will be asked if she intends to check her skin again. In addition, she will be asked if she intends to check the skin of family members. Women will be invited to take a brochure to help implement SSE.

The screening questions are as follows:

1. During your visit for mammography, did you notice any information about checking your skin for melanoma?

   ___Yes __ No
2. Did you think this applied to you? ___Yes __ No
3. If no, why not? (open ended)
4. If yes, why? (open ended)
5. Did you check your skin? (If no, please proceed to question #8)

   ___Yes __ No
6. If yes, did you notice any concerning moles?

   * Yes __ No
7. If yes, may we contact you by telephone or email in 2 weeks to see if you have made an appointment to see a dermatologist?

   ___Yes __ No If yes, which way do you prefer to be contacted?

   Phone _________________________(Number) Email _________________________ (Address)
8. If no, will you consider checking your skin in the future?

   ___Yes __ No
9. If yes, may we contact you by telephone or email in 2 weeks to see if you have checked your skin for any concerning moles?

   ___Yes __ No If yes, which way do you prefer to be contacted?

   Phone _________________________(Number) Email _________________________ (Address)
10. If you found any concerning moles, did you make an appointment to see a dermatologist.

    * Yes __ No

The RA will record the responses. Women who checked their skin ,either today or in about 2 weeks, will be invited to participate in a survey about skin location(s) checked, use of the SSE kit, and their decision about the spot on the skin.

ELIGIBILITY:
Inclusion Criteria:

- Qualitative research: structured interview Women 18 years of age and older, who are waiting to have a mammogram Women agree to a structured interview regarding knowledge of melanoma and awareness of melanoma risk.

Following development of a draft of a brochure, women will agree to review a draft and provide comment during a 5 minute interview

* Qualitative research: focus group Women 18 years of age and older Women with a history of regular mammograms Women with a history of indoor tanning, a personal history of skin cancer, and/or a family history of skin cancer Women willing to participate in a 60 minute focus group to assess materials to be provided during the mammogram experience
* Quantitative research

Women 18 years of age and older who respond positively to the three screening questions:

Noticed information about checking your skin for melanoma. Thought this information was applicable to them. Checked skin or will consider checking skin in the future.

Exclusion Criteria:

* Women who are unable to see to read a newspaper, unable to read English, and who have cognitive impairment causing problems with functioning at a sixth grade reading level or inability to speak.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 560 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Performance of SSE | 4 weeks
  Checked Moles

SECONDARY OUTCOMES:
Questionnaire to identify concerning moles | 2 weeks
  Found Concerning mole

OTHER OUTCOMES:
Management of decision | 2 weeks
  Made appointment to see a doctor about the mole

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No